CLINICAL TRIAL: NCT00888069
Title: A Randomized, Open-Label, Single-Dose Pilot Study of Oral and i.v. CTAP101 Evaluating PK and Safety in Stage 3 and 4 CKD Subjects With Vitamin D Insufficiency and SHPT
Brief Title: Pharmacokinetics and Safety Pilot Study of Single-Dose Oral and Intravenous CTAP101 in Stage 3 and 4 Chronic Kidney Disease Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO IP Holdings II, Inc. (Industry)
Responsible Party: Sponsor
Organization: OPKO Health, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTAP101-CL-2004
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism; Chronic Renal Insufficiency; Chronic Renal Failure
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Renal Insufficiency, Chronic; Kidney Diseases; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Kidney Failure, Chronic; Parathyroid Diseases; Renal Insufficiency; Hyperparathyroidism; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose CTAP101 Capsules (Experimental): CTAP101 Capsules, 450 mcg dose
  Interventions: Drug: CTAP101 Capsules
- High Dose CTAP101 Capsules (Experimental): CTAP101 Capsules, 900 mcg dose
  Interventions: Drug: CTAP101 Capsules
- CTAP101 Injection (Experimental): IV injection, 448 mcg dose
  Interventions: Drug: CTAP101 Injection

INTERVENTIONS:
Drug: CTAP101 Capsules — Single dose oral administration
  Arms: High Dose CTAP101 Capsules; Low Dose CTAP101 Capsules
Drug: CTAP101 Injection — single IV injection
  Arms: CTAP101 Injection

SUMMARY:
This study will investigate how the levels of a single dose of CTAP101 changes in the body over time (pharmacokinetics, PK) and how CTAP101 affects other mineral and hormonal balances (pharmacodynamics, PD) in patients with Stage 3 or 4 chronic kidney disease (CKD) with vitamin D insufficiency and secondary hyperparathyroidism (SHPT).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between great than or equal to 18 and less than or equal to 40 kg/m2
* Plasma iPTH value for Stage 3 CKD greater than or equal to 70 pg/mL and lower than or equal to 1000 pg/mL
* Plasma iPTH value for Stage 4 CKD greater than or equal to 110 pg/mL and lower than or equal to 1000 pg/mL
* Adjusted serum total calcium value greater than 8.4 mg/dL and lower than 10.0 mg/dL
* Serum phosphorus value greater than or equal to 2.5 mg/dL and lower than or equal to 5.5 mg/dL
* Serum 25-hydroxyvitamin D level greater than 15 ng/mL and lower than 30 ng/mL
* Hemoglobin level greater than or equal to 10 g/dL

Exclusion Criteria:

* Has nephrotic range proteinuria
* Has liver disease or significant hepatic dysfunction
* Is taking Cytochrome P450 3A4 inhibitors or inducers
* Has adult history of kidney stones and dysphagia
* Has known history of alcohol/controlled substance abuse or are positive for drug of abuse screen
* Currently on dialysis
* Current serious illness such as cancer, HIV, cardiovascular event or hepatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the PK and bioavailability of CTAP101 in Stage 3 and 4 CKD subjects with vitamin D insufficiency and SHPT | from 3 to 0 hours prior to dosing until 42 days post dosing

SECONDARY OUTCOMES:
To assess the safety and tolerability of CTAP101 capsules and injection | From signing of ICF (Day -35) through study completion (Day 42 post dosing)
To assess the pharmacodynamics of single dose CTAP101 in Stage 3 and Stage 4 CKD subjects with vitamin D insufficiency and SHPT. | From signing of ICF (Day -35) through study completion (Day 42 post dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Renal
Locations (12):
- United States (12):
  - Pivotal Research Centers, Peoria, Arizona
  - Research by Design, Evergreen Park, Illinois
  - Western New England Renal & Transplant Associates, Springfield, Massachusetts
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - DCI, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Northeast Clinical Research, Allentown, Pennsylvania
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Southwest Houston Research Ltd, Houston, Texas
  - Purity Dialysis Centers / Nephrology Associates, Delafield, Wisconsin
  - Gunderson Clinic Ltd., La Crosse, Wisconsin